CLINICAL TRIAL: NCT01981577
Title: Ultra-high Field Imaging of the Cortico-striato-subthalamic Functional and Structural Connectivity to Improve Deep Brain Stimulation Surgery in Parkinson's Disease Patients
Brief Title: Subthalamic Nucleus Connectivity in Parkinson's Disease With Ultra-high Field Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: NL42613.068.13
Record Dates: First submitted 2013-09-30; First posted 2013-11-11 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Subthalamic Nucleus; Ultrahigh field Magnetic Resonance imaging; Functional connectivity; Structural connectivity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Patients with Parkinson's Disease
- Healthy volunteers

SUMMARY:
The purpose of this study is to investigate the segregation of the subthalamic nucleus into its motor and non-motor regions in patients with Parkinson's disease and healthy controls with the aid of ultra-high field magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

Both groups:

* Mental competence

Group 1:

* Parkinson's disease patients scheduled for deep brain stimulation surgery

Group 2:

* Age and gender matched volunteers

Exclusion Criteria:

Both groups:

* Head injury
* Stroke
* Other neurological diseases other than Parkinson's disease
* Metallic prostheses or pacemaker in the subject's body or other contra indications for MRI

Group 1:

* Inability to abstain from dopaminergic drug use

Group 2:

* Parkinson's disease
* Use of medication affecting the central nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Parkinson's patients scheduled for deep brain stimulation surgery at Maastricht University Medical Center
  * Healthy volunteers from a community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Voxels of the subthalamic nucleus that are structurally or functionally connected to the motor cortex. | One measurement, consisting of 1 MRI scan of 1 hour
  Two brain areas are said to be structurally connected if they are connected by fiber tracks computed from diffusion weighted MRI data.
  Two brain areas are said to be functionally connected if they show statistically significantly correlated resting state functional MRI signals.

SECONDARY OUTCOMES:
Strength of the structural and functional connectivity between the subthalamic nucleus and the motor cortex. | One measurement, consisting of 1 MRI scan of 1 hour
  Strength of the structural connectivity is defined as: fractional anisotropy along computed fiber tracks between the subthalamic nucleus and the motor cortex.
  Strength of the functional connectivity is defined as: height of the correlation between the resting state functional MRI signals in the subthalamic nucleus and the motor cortex.
Brain areas structurally and functionally connected to the stimulation zone of the optimal electrode of operated Parkinson's patients. | One measurement, consisting of 1 MRI scan of 1 hour
  This results in a list with brain structures that are functionally and/or structurally connected to the stimulation zone.
Brain areas that show an activation pattern measured with functional magnetic resonance imaging, that is correlated to a motor task. | One measurement, consisting of 1 MRI scan of 1 hour
  This results in a list of brain areas that are related to the motor task.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Temel, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands